CLINICAL TRIAL: NCT01843335
Title: Contrast-enhanced Ultrasound in Follow-up After Endovascular Aneurysm Repair
Status: Terminated | Type: Observational
Why Stopped: recruitment too slow
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); SINTEF Health Research (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/359/REKnord
Record Dates: First submitted 2013-04-26; First posted 2013-04-30 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Abdominal Aortic Aneurysm; Endoleak
Keywords: Cardiovascular Diagnostic Technique; Ultrasound
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Endoleak

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
X-ray computed tomography imaging (CT) is routinely used in follow-up after endovascular aneurysm repair (EVAR). Contrast-enhanced ultrasound (CEUS) has been shown to give accurate information about endoleak after EVAR. Benefits of CEUS over CT include less radiation exposure, avoidance of renal function deterioration due to repeated X-ray contrast agent application and decrease in the cost of EVAR follow-up. This study is designed to investigate if results from literature are reproducible in St Olavs Hospital in Trondheim (Norway), to gain experience with the technique and to introduce CEUS as an alternative for detection of endoleak in this hospital.

ELIGIBILITY:
Inclusion Criteria:

* in follow-up after endovascular implantation of abdominal aortic prothesis

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients in follow-up after endovascular implantation of abdominal aortic prothesis, Central Norway
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Detection of endoleak with CEUS | 9 months
  Compare CEUS with computed tomography angiography (CTA) sensitivity for detection of endoleak

CONTACTS AND LOCATIONS:
Overall Officials: Reidar Brekken, PhD, Study Director — National Taiwan Normal University
Locations (1):
- St Olavs Hospital, Trondheim, Norway